CLINICAL TRIAL: NCT00934037
Title: Multi Center Combined Non-invasive Coronary Angiography and Myocardial Perfusion Imaging Using 320-Detector Computed Tomography
Brief Title: Combined Non-invasive Coronary Angiography and Myocardial Perfusion Imaging Using 320 Detector Computed Tomography
Acronym: Core320
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Toshiba America Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: NA_00022661; Core320 (Other: Other)
Record Dates: First submitted 2009-05-11; First posted 2009-07-08 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Arterial Occlusive Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia; Vascular Diseases; Arteriosclerosis; Ischemia; Coronary Artery Disease
Keywords: Coronary Artery Disease; Computed Tomography; Myoperfusion; Angiography; SPECT
MeSH Terms: conditions — Arterial Occlusive Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia; Vascular Diseases; Arteriosclerosis; Ischemia; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined CT Angiography and Myocardial Perfusion (Other): Single Arm study. All patients underwent combined CT Angiography and Myocardial Perfusion.
  Interventions: Procedure: 320 Volume Detector Computed Tomography; Other: Other: Multidetector Computed Tomography - 320 detectors

INTERVENTIONS:
Procedure: 320 Volume Detector Computed Tomography — Single Arm Study. All patients undergo Volume (Multidetector) CT.
Other: Other: Multidetector Computed Tomography - 320 detectors — Multidetector computed tomography angiography
  Other Names: Aquilion ONE CT scanner

SUMMARY:
The purpose of this study is to evaluate the diagnostic accuracy of multi-detector computed tomography using 320 detectors for identifying the combination of coronary artery stenosis ≥ 50% and a corresponding myocardium perfusion defect in a patient with suspected coronary artery disease compared with conventional coronary angiography and single photon emission computed tomography myocardium perfusion imaging.

DETAILED DESCRIPTION:
The Combined Coronary angiography and myocardial perfusion imaging using 320 detectors computed tomography (CORE-320) was designed as a prospective, multi-center, international, blinded study designed to evaluate the diagnostic accuracy of multi-detector computed tomography using 320 detectors for identifying coronary artery luminal stenosis and corresponding myocardium perfusion defects in patients with suspected coronary artery disease. The primary analysis will be a comparison of the diagnostic capability of the combination of quantitative 320-MDCT angiography and quantitative perfusion imaging to the combination of conventional coronary angiography and SPECT myocardial perfusion imaging at the patient level. A positive patient will be defined as having at least one vessel with a ≥ 50% diameter stenosis defined by quantitative coronary angiography and a corresponding positive SPECT territorial myocardial perfusion defect.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age 45-85. Women of child bearing potential must demonstrate a negative pregnancy test within 24 hours of the study MDCT.
* Suspected or diagnosed coronary artery disease with a clinical indication for coronary angiography; and planned coronary angiography within the next 60 days.
* Able to understand and willing to sign the Informed Consent Form.

Exclusion Criteria:

* Known allergy to iodinated contrast media.
* History of contrast-induced nephropathy.
* History of multiple myeloma or previous organ transplantation.
* Elevated serum creatinine (> 1.5 mg/dl) OR calculated creatinine clearance of < 60 ml/min (using the Cockcroft-Gault formula.
* Atrial fibrillation or uncontrolled tachyarrhythmia, or advanced atrioventricular block (second or third degree heart block).
* Evidence of severe symptomatic heart failure (NYHA Class III or IV); Known or suspected moderate or severe aortic stenosis.
* Previous coronary artery bypass or other cardiac surgery.
* Coronary artery intervention within the last 6 months.
* Known or suspected intolerance or contraindication to beta-blockers including:

  * Known allergy to beta-blockers
  * History of moderate to severe bronchospastic lung disease (including moderate to severe asthma).
* Severe pulmonary disease (chronic obstructive pulmonary disease).
* Presence of any other history or condition that the investigator feels would be problematic.
* SPECT preformed in non-validated center within 60 days prior to screening.
* SPECT performed within the previous 6 months of screening but > 60 days.
* SPECT studies performed within 60 days of screening that include rest and stress studies performed using 2 day protocols.
* BMI greater than 40

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of volume (multi-detector) computed tomography using 320 detectors in a patient with suspected coronary artery disease. | 30-60 Days
  Diagnostic accuracy of volume (multi-detector) computed tomography using 320 detectors for identifying coronary artery luminal stenosis and corresponding myocardium perfusion defects in a patient with suspected coronary artery disease.

SECONDARY OUTCOMES:
Diagnostic accuracy of volume computed tomography using 320 detectors in a vessel of a patient with suspected coronary artery disease. | 30-60 Days
  Diagnostic accuracy of volume computed tomography using 320 detectors for identifying coronary artery luminal stenosis and corresponding territorial myocardium perfusion defects in a vessel of a patient with suspected coronary artery disease.
Compare the relative diagnostic accuracy of 320 CT angiography vs SPECT in predicting at least one ≥ 50% coronary stenosis detected by QCA | 30-60 Days
  Compare the relative diagnostic accuracy of 320 CT angiography vs SPECT in predicting at least one ≥ 50% coronary stenosis detected by QCA
Compare the relative diagnostic accuracy of 320 CT perfusion vs SPECT in predicting at least one ≥ 50% coronary stenosis detected by quantitative conventional angiography. | 30-60 Days
  Compare the relative diagnostic accuracy of 320 CT perfusion vs SPECT in predicting at least one ≥ 50% coronary stenosis detected by quantitative conventional angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Joao AC Lima, MD MBA, Study Chair — Johns Hopkins School of Medicine
Locations (16):
- United States (4):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - National Heart Lung and Blood Institute (NHLBI), Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women Hospital, Boston, Massachusetts
- Brazil (2):
  - Albert Einstein Hospital, São Paulo
  - INCOR Heart Institute University-Sao Paulo, São Paulo
- Toronto General Hospital, Toronto, Canada
- Rigshospitalet - University of Copenhagen, Blegdamsvej, Denmark
- Charite Humboldt University, Berlin, Germany
- Japan (4):
  - Iwate Medical University, Morioka
  - Keio University, Tokyo
  - St. Luke's International Hospital, Tokyo
  - Mie University, Tsu
- Leiden University, Leiden, Netherlands
- Singapore (2):
  - Mount Elizabeth Hospital, Singapore
  - National Heart Center, Singapore

REFERENCES:
- [Background] Miller JM, Rochitte CE, Dewey M, Arbab-Zadeh A, Niinuma H, Gottlieb I, Paul N, Clouse ME, Shapiro EP, Hoe J, Lardo AC, Bush DE, de Roos A, Cox C, Brinker J, Lima JA. Diagnostic performance of coronary angiography by 64-row CT. N Engl J Med. 2008 Nov 27;359(22):2324-36. doi: 10.1056/NEJMoa0806576. PMID 19038879
- [Background] Vavere AL, Simon GG, George RT, Rochitte CE, Arai AE, Miller JM, Di Carli M, Arbab-Zadeh A, Dewey M, Niinuma H, Laham R, Rybicki FJ, Schuijf JD, Paul N, Hoe J, Kuribyashi S, Sakuma H, Nomura C, Yaw TS, Kofoed KF, Yoshioka K, Clouse ME, Brinker J, Cox C, Lima JA. Diagnostic performance of combined noninvasive coronary angiography and myocardial perfusion imaging using 320 row detector computed tomography: design and implementation of the CORE320 multicenter, multinational diagnostic study. J Cardiovasc Comput Tomogr. 2011 Nov-Dec;5(6):370-81. doi: 10.1016/j.jcct.2011.11.001. Epub 2011 Nov 12. PMID 22146496
- [Background] Miller JM, Dewey M, Vavere AL, Rochitte CE, Niinuma H, Arbab-Zadeh A, Paul N, Hoe J, de Roos A, Yoshioka K, Lemos PA, Bush DE, Lardo AC, Texter J, Brinker J, Cox C, Clouse ME, Lima JA. Coronary CT angiography using 64 detector rows: methods and design of the multi-centre trial CORE-64. Eur Radiol. 2009 Apr;19(4):816-28. doi: 10.1007/s00330-008-1203-7. Epub 2008 Nov 8. PMID 18998142
- [Background] Yoneyama K, Vavere AL, Cerci R, Ahmed R, Arai AE, Niinuma H, Rybicki FJ, Rochitte CE, Clouse ME, George RT, Lima JA, Arbab-Zadeh A. Influence of image acquisition settings on radiation dose and image quality in coronary angiography by 320-detector volume computed tomography: the CORE320 pilot experience. Heart Int. 2012 Jun 5;7(2):e11. doi: 10.4081/hi.2012.e11. Epub 2012 Jun 25. PMID 23185678
- [Background] Cerci RJ, Arbab-Zadeh A, George RT, Miller JM, Vavere AL, Mehra V, Yoneyama K, Texter J, Foster C, Guo W, Cox C, Brinker J, Di Carli M, Lima JA. Aligning coronary anatomy and myocardial perfusion territories: an algorithm for the CORE320 multicenter study. Circ Cardiovasc Imaging. 2012 Sep 1;5(5):587-95. doi: 10.1161/CIRCIMAGING.111.970608. Epub 2012 Aug 10. PMID 22887690
- [Background] George RT, Arbab-Zadeh A, Miller JM, Vavere AL, Bengel FM, Lardo AC, Lima JA. Computed tomography myocardial perfusion imaging with 320-row detector computed tomography accurately detects myocardial ischemia in patients with obstructive coronary artery disease. Circ Cardiovasc Imaging. 2012 May 1;5(3):333-40. doi: 10.1161/CIRCIMAGING.111.969303. Epub 2012 Mar 23. PMID 22447807
- [Background] George RT, Arbab-Zadeh A, Cerci RJ, Vavere AL, Kitagawa K, Dewey M, Rochitte CE, Arai AE, Paul N, Rybicki FJ, Lardo AC, Clouse ME, Lima JA. Diagnostic performance of combined noninvasive coronary angiography and myocardial perfusion imaging using 320-MDCT: the CT angiography and perfusion methods of the CORE320 multicenter multinational diagnostic study. AJR Am J Roentgenol. 2011 Oct;197(4):829-37. doi: 10.2214/AJR.10.5689. PMID 21940569
- [Background] Mehra VC, Valdiviezo C, Arbab-Zadeh A, Ko BS, Seneviratne SK, Cerci R, Lima JA, George RT. A stepwise approach to the visual interpretation of CT-based myocardial perfusion. J Cardiovasc Comput Tomogr. 2011 Nov-Dec;5(6):357-69. doi: 10.1016/j.jcct.2011.10.010. Epub 2011 Oct 31. PMID 22146495
- [Derived] Preuss D, Garcia G, Laule M, Dewey M, Rief M. Myocardial CT perfusion imaging for the detection of obstructive coronary artery disease: multisegment reconstruction does not improve diagnostic performance. Eur Radiol Exp. 2022 Jan 31;6(1):5. doi: 10.1186/s41747-021-00256-8. PMID 35099638
- [Derived] Dewey M, Rochitte CE, Ostovaneh MR, Chen MY, George RT, Niinuma H, Kitagawa K, Laham R, Kofoed K, Nomura C, Sakuma H, Yoshioka K, Mehra VC, Jinzaki M, Kuribayashi S, Laule M, Paul N, Scholte AJ, Cerci R, Hoe J, Tan SY, Rybicki FJ, Matheson MB, Vavere AL, Arai AE, Miller JM, Cox C, Brinker J, Clouse ME, Di Carli M, Lima JAC, Arbab-Zadeh A. Prognostic value of noninvasive combined anatomic/functional assessment by cardiac CT in patients with suspected coronary artery disease - Comparison with invasive coronary angiography and nuclear myocardial perfusion imaging for the five-year-follow up of the CORE320 multicenter study. J Cardiovasc Comput Tomogr. 2021 Nov-Dec;15(6):485-491. doi: 10.1016/j.jcct.2021.04.005. Epub 2021 May 12. PMID 34024757
- [Derived] Kishi S, Magalhaes TA, Cerci RJ, Zimmermann E, Matheson MB, Vavere A, Tanami Y, Kitslaar PH, George RT, Brinker J, Miller JM, Clouse ME, Lemos PA, Niinuma H, Reiber JHC, Kofoed KF, Rochitte CE, Rybicki FJ, Di Carli MF, Cox C, Lima JAC, Arbab-Zadeh A. Comparative effectiveness of coronary artery stenosis and atherosclerotic plaque burden assessment for predicting 30-day revascularization and 2-year major adverse cardiac events. Int J Cardiovasc Imaging. 2020 Dec;36(12):2365-2375. doi: 10.1007/s10554-020-01851-3. Epub 2020 May 2. PMID 32361925
- [Derived] Schuijf JD, Matheson MB, Ostovaneh MR, Arbab-Zadeh A, Kofoed KF, Scholte AJHA, Dewey M, Steveson C, Rochitte CE, Yoshioka K, Cox C, Di Carli MF, Lima JAC. Ischemia and No Obstructive Stenosis (INOCA) at CT Angiography, CT Myocardial Perfusion, Invasive Coronary Angiography, and SPECT: The CORE320 Study. Radiology. 2020 Jan;294(1):61-73. doi: 10.1148/radiol.2019190978. Epub 2019 Nov 19. PMID 31746688
- [Derived] Song YB, Arbab-Zadeh A, Matheson MB, Ostovaneh MR, Vavere AL, Dewey M, Rochitte C, Niinuma H, Laham R, Schuijf JD, Cox C, Brinker J, di Carli M, Lima JAC, Miller JM. Contemporary Discrepancies of Stenosis Assessment by Computed Tomography and Invasive Coronary Angiography. Circ Cardiovasc Imaging. 2019 Feb;12(2):e007720. doi: 10.1161/CIRCIMAGING.118.007720. PMID 30764641
- [Derived] Rief M, Chen MY, Vavere AL, Kendziora B, Miller JM, Bandettini WP, Cox C, George RT, Lima J, Di Carli M, Plotkin M, Zimmermann E, Laule M, Schlattmann P, Arai AE, Dewey M. Coronary Artery Disease: Analysis of Diagnostic Performance of CT Perfusion and MR Perfusion Imaging in Comparison with Quantitative Coronary Angiography and SPECT-Multicenter Prospective Trial. Radiology. 2018 Feb;286(2):461-470. doi: 10.1148/radiol.2017162447. Epub 2017 Sep 25. PMID 28956734
- [Derived] Penagaluri A, Higgins AY, Vavere AL, Miller JM, Arbab-Zadeh A, Betoko A, Steveson C, Zimmermann E, Cox C, Rochitte CE, Dewey M, Kofoed KF, Niinuma H, Di Carli MF, Lima JA, Chen MY. Computed Tomographic Perfusion Improves Diagnostic Power of Coronary Computed Tomographic Angiography in Women: Analysis of the CORE320 Trial (Coronary Artery Evaluation Using 320-Row Multidetector Computed Tomography Angiography and Myocardial Perfusion) According to Gender. Circ Cardiovasc Imaging. 2016 Nov;9(11):e005189. doi: 10.1161/CIRCIMAGING.116.005189. PMID 27811151
- [Derived] Arbab-Zadeh A, Di Carli MF, Cerci R, George RT, Chen MY, Dewey M, Niinuma H, Vavere AL, Betoko A, Plotkin M, Cox C, Clouse ME, Arai AE, Rochitte CE, Lima JA, Brinker J, Miller JM. Accuracy of Computed Tomographic Angiography and Single-Photon Emission Computed Tomography-Acquired Myocardial Perfusion Imaging for the Diagnosis of Coronary Artery Disease. Circ Cardiovasc Imaging. 2015 Oct;8(10):e003533. doi: 10.1161/CIRCIMAGING.115.003533. PMID 26467105
- [Derived] Sharma RK, Arbab-Zadeh A, Kishi S, Chen MY, Magalhaes TA, George RT, Dewey M, Rybicki FJ, Kofoed KF, de Roos A, Tan SY, Matheson M, Vavere A, Cox C, Clouse ME, Miller JM, Brinker JA, Arai AE, Di Carli MF, Rochitte CE, Lima JA. Incremental diagnostic accuracy of computed tomography myocardial perfusion imaging over coronary angiography stratified by pre-test probability of coronary artery disease and severity of coronary artery calcification: The CORE320 study. Int J Cardiol. 2015 Dec 15;201:570-7. doi: 10.1016/j.ijcard.2015.05.110. Epub 2015 May 19. PMID 26334382
- [Derived] Magalhaes TA, Kishi S, George RT, Arbab-Zadeh A, Vavere AL, Cox C, Matheson MB, Miller JM, Brinker J, Di Carli M, Rybicki FJ, Rochitte CE, Clouse ME, Lima JA. Combined coronary angiography and myocardial perfusion by computed tomography in the identification of flow-limiting stenosis - The CORE320 study: An integrated analysis of CT coronary angiography and myocardial perfusion. J Cardiovasc Comput Tomogr. 2015 Sep-Oct;9(5):438-45. doi: 10.1016/j.jcct.2015.03.004. Epub 2015 Mar 21. PMID 25977111
- [Derived] Rybicki FJ, Mather RT, Kumamaru KK, Brinker J, Chen MY, Cox C, Matheson MB, Dewey M, DiCarli MF, Miller JM, Geleijns J, George RT, Paul N, Texter J, Vavere A, Yaw TS, Lima JA, Clouse ME. Comprehensive assessment of radiation dose estimates for the CORE320 study. AJR Am J Roentgenol. 2015 Jan;204(1):W27-36. doi: 10.2214/AJR.13.12375. PMID 25539270